CLINICAL TRIAL: NCT01712178
Title: Study to Assess the Pharmacokinetic, Pharmacodynamic, Safety and Immunogenicity of a New Adalimumab Formulation in Subjects With Active Rheumatoid Arthritis
Brief Title: A Study in Rheumatoid Arthritis (RA) Patients to Compare Two Formulations of Adalimumab for Pharmacokinetic, Pharmacodynamic and Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-390; 2012-000535-36 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-10-23 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Pharmacodynamic,Pharmacokinetic
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New formulation of adalimumab 40 mg every other week (Experimental): New formulation adalimumab 40 mg every other week
  Interventions: Biological: Adalimumab, new formulation
- Current formulation adalimumab 40 mg every other week (Active Comparator): Current formulation adalimumab 40 mg every other week
  Interventions: Biological: Adalimumab, current formulation

INTERVENTIONS:
Biological: Adalimumab, current formulation — Current formulation adalimumab 40 mg every other week
  Other Names: Humira
  Arms: Current formulation adalimumab 40 mg every other week
Biological: Adalimumab, new formulation — New formulation adalimumab 40 mg every other week
  Arms: New formulation of adalimumab 40 mg every other week

SUMMARY:
A study in Rheumatoid Arthritis (RA) patients to evaluate two formulations of adalimumab for pharmacodynamics, pharmacokinetics, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, 18 years or older who has a diagnosis of Rheumatoid Arthritis (RA) as defined by the 1987-revised American College of Rheumatology (ACR)-classification criteria or the new American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) diagnostic criteria for RA 2010-classification criteria and has a disease duration for a minimum of 3 months.
* Subjects must be naïve to biologic therapy.
* Subject must meet the following criteria for the joint assessment: • At least 6 swollen joints out of 66 assessed. • At least 6 tender joints out of 68 assessed.
* Prior Disease Modifying Antirheumatic Drug (DMARD) therapy: a) Subjects not on methotrexate at baseline must remain without methotrexate throughout the study. Subjects on prior Methotrexate (MTX) must have discontinued at least 28 days prior to Week 0 (Day 1). b) Subjects on Disease Modifying Antirheumatic Drug (DMARD) therapy other than Methotrexate (MTX) (except prednisone/prednisolone less than or equal to 10 mg) must discontinue it for at least 28 days before the first dose of investigational product at Week 0 (Day 1).
* Female subjects are either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy), or are practicing at least 1 of the following methods of birth control throughout the study and for at least 150 days after the last dose of study drug: • Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD). • Hormonal contraceptives for 90 days prior to study drug administration. • Vasectomized partner(s).
* Subjects must be able and willing to self-administer subcutaneous (SC) injections or have a qualified person available to administer subcutaneous (SC) injections.
* Subject is judged to be in good general health as determined by the Principal Investigator based upon the results of medical history, physical examination, laboratory profile, chest x-ray (CXR), and 12 lead electrocardiogram (ECG) performed during Screening.
* Subject has a negative Tuberculosis (TB) screening assessment (including a (Purified Protein Derivative (PPD) test or QuantiFERON-Tuberculosis (TB) Gold test or equivalent) and negative chest x-ray (Posterior-Anterior (PA) and lateral view) at Screening. If a subject has evidence of a latent Tuberculosis (TB) infection, the subject must initiate and complete a minimum of 2 weeks of anti-Tuberculosis (TB) therapy or have documented completion of a course of anti-Tuberculosis (TB) therapy prior to Baseline.
* Subjects must be willing to provide written consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

* Subject has been treated with intra-articular or parenteral administration of corticosteroids in the preceding 4 weeks from Baseline visit. Inhaled corticosteroids for stable medical conditions are allowed. Oral of less than or equal to 10 mg/d prednisone equivalent are allowed.
* Subject has been treated with any investigational drug of a chemical or biological nature within a minimum of 30 days or 5 half-lives (whichever is longer) of the drug prior to Baseline Visit.
* Subject has a history of acute inflammatory joint disease of different origin other than Rheumatoid Arthritis (RA) (e.g., seronegative spondyloarthropathy, psoriatic arthritis, Reiter's syndrome, systemic lupus erythematosus, gouty arthritis, or any arthritis with onset prior to age 17 years).
* Known hypersensitivity to adalimumab or its excipients.
* Subject currently uses or plans to use anti-retroviral therapy at any time during the study.
* History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
* History of invasive infection (e.g., listeriosis and histoplasmosis), human immunodeficiency syndrome (HIV).
* Chronic recurring infections or active Tuberculosis (TB).
* History of moderate to severe congestive heart failure (New York Heart Association (NYHA) class III or IV), recent cerebrovascular accident and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
* Subject received any live vaccine within 3 months prior to study drug administration. - Subject has a history of clinically significant hematologic (e.g., severe anemia, leukopenia, thrombocytopenia), renal or liver disease (e.g., fibrosis, cirrhosis, hepatitis).
* Positive pregnancy test at Screening or Baseline.
* Subject is considered by the investigator, for any reason, to be unsuitable candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Payne, PhD, Study Director — AbbVie
Locations (21):
- United States (6):
  - Site Reference ID/Investigator# 75073, Mesa, Arizona
  - Site Reference ID/Investigator# 75077, Hemet, California
  - Site Reference ID/Investigator# 75076, Wichita, Kansas
  - Site Reference ID/Investigator# 75075, Clifton, New Jersey
  - Site Reference ID/Investigator# 83133, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 75074, Charleston, South Carolina
- Belgium (2):
  - Site Reference ID/Investigator# 75100, Brussels
  - Site Reference ID/Investigator# 75101, Liège
- Czechia (4):
  - Site Reference ID/Investigator# 75104, Brno
  - Site Reference ID/Investigator# 76788, Prague
  - Site Reference ID/Investigator# 75102, Uherské Hradiště
  - Site Reference ID/Investigator# 75103, Zlín
- Site Reference ID/Investigator# 78014, Ratingen, Germany
- Puerto Rico (2):
  - Site Reference ID/Investigator# 75079, Caguas
  - Site Reference ID/Investigator# 75078, Vega Baja
- Romania (3):
  - Site Reference ID/Investigator# 76787, Bucharest
  - Site Reference ID/Investigator# 75978, Cluj-Napoca
  - Site Reference ID/Investigator# 76433, Ploieşti
- Slovakia (3):
  - Site Reference ID/Investigator# 76934, Banská Bystrica
  - Site Reference ID/Investigator# 76935, Senica
  - Site Reference ID/Investigator# 76682, Žilina

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US prescribing information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Started | 50 | 50
Completed | 49 | 47
Not Completed | 1 | 3
Not completed — Withdrew consent due to an adverse event | 1 | 1
Not completed — Serious adverse event/withdrew consent | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.0) | 53.0 (12.3) | 54.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentrations of Adalimumab at Weeks 12 and 24
Description: Blood samples for adalimumab analysis were collected by venipuncture and serum concentrations of adalimumab were determined using a validated enzyme-linked immunoadsorbent assay (ELISA) method.
Time Frame: Measured at Weeks 12 and 24
Population: Data from participants receiving the new formulation of adalimumab were analyzed for 46 and 47 participants, respectively, at weeks 12 and 24. Data for the participants receiving the current formulation of adalimumab were analyzed for 43 participants at week 12 and 41 participants at week 24.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 47 | 43
µg/mL
  Week 12: n= 46 (new), n=43 (current) | 5.72 (4.49) | 6.23 (4.29)
  Week 24: n= 47 (new), n=41 (current) | 5.95 (5.13) | 6.17 (4.50)

2. Primary Outcome: Mean Disease Activity Scores (DAS28) at Weeks 12 and 24
Description: The Disease Activity Score (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Measured at Weeks 12 and 24
Population: All available data were included. If a subject did not have a value for a given time of evaluation, but did have a value at times previous to this after the study drug treatment began, the last available value was used to replace the missing value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 50
units on a scale
  Week 12 | 3.78 (0.147) | 3.82 (0.148)
  Week 24 | 3.54 (0.152) | 3.46 (0.153)

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Weeks 12 and 24
Description: American College of Rheumatology 20% (ACR20) response. A participant is a responder if the following 3 criteria for improvement from baseline are met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment Questionnaire
    * CRP (Acute phase reactant (Erythrocyte sedimentation rate/C-reactive protein))
Time Frame: Measured at Weeks 12 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 50
percentage of participants
  Week 12 | 62.0 | 68.0
  Week 24 | 68.0 | 68.0

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response at Weeks 12 and 24
Description: American College of Rheumatology 50% (ACR50) response. A participant is a responder if the following 3 criteria for improvement from baseline are met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment Questionnaire
    * CRP (Acute phase reactant (Erythrocyte sedimentation rate/C-reactive protein))
Time Frame: Measured at Weeks 12 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 50
percentage of participants
  Week 12 | 36.0 | 40.0
  Week 24 | 48.0 | 50.0

5. Secondary Outcome: Mean Health Assessment Questionnaire (HAQ-DI) Scores at Weeks 12 and 24
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥0.22. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5.
Time Frame: Measured at Weeks 12 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 50
units on a scale
  Week 12 | 1.10 (0.075) | 1.02 (0.076)
  Week 24 | 1.01 (0.082) | 0.97 (0.083)

6. Secondary Outcome: Mean Short Form-36 (SF-36) Physical Component Summary Scores and Mental Component Summary Scores at Weeks 12 and 24
Description: The Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 (maximum disability) - 100 (no disability). The standard recall period is four weeks.
Time Frame: Measured at Weeks 12 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 49
units on a scale
  PCS score- Week 12 | 38.88 (0.957) | 39.08 (0.974)
  PCS score- Week 24 | 39.38 (1.044) | 39.94 (1.022)
  MCS score- Week 12 | 44.78 (1.172) | 42.78 (1.192)
  MCS score- Week 24 | 43.16 (1.246) | 45.46 (1.267)

7. Secondary Outcome: Percentage of Participants Positive for Anti-adalimumab Antibody
Description: Percentage of participants with anti-adalimumab antibody
Time Frame: Measured through Week 24
Measure: Number; unit: Percentage of participants
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 50
Percentage of participants | 14 | 16

8. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. See the Reported Adverse Events Section for more details.
Time Frame: From time of informed consent to 70 days following the last dose of study drug
Measure: Number; unit: participants
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 50 | 50
participants | 31 | 34

9. Secondary Outcome: Mean Injection Site Pain on a Visual Analogue Scale (VAS)
Description: The Visual Analogue Scale (VAS) consisted of a horizontal 100 mm line, with 0 representing "no pain" and 100 representing "worst possible pain". Participants placed a mark on the line representing their current level of pain immediately after injections on Day 1 of the study.
Time Frame: Immediately after injections on Day 1
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 49 | 50
Millimeters | 14.4 (22.6) | 35.9 (29.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 70 days following the last dose. Serious adverse events were collected from the time the participant signed the informed consent.
Arm/Group | New Formulation of Adalimumab 40 mg Every Other Week | Current Formulation Adalimumab 40 mg Every Other Week
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/50
Other Adverse Events (participants affected / at risk) | 23/50 | 16/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Formulation of Adalimumab 40 mg Every Other Week (N=50) | Current Formulation Adalimumab 40 mg Every Other Week (N=50)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Formulation of Adalimumab 40 mg Every Other Week (N=50) | Current Formulation Adalimumab 40 mg Every Other Week (N=50)
DYSPEPSIA (Gastrointestinal disorders) | 3 | 1
NAUSEA (Gastrointestinal disorders) | 4 | 0
INJECTION SITE REACTION (General disorders) | 3 | 0
CYSTITIS (Infections and infestations) | 4 | 2
NASOPHARYNGITIS (Infections and infestations) | 5 | 6
SINUSITIS (Infections and infestations) | 3 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 4
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.